CLINICAL TRIAL: NCT02009735
Title: Virosensor -Based Real-time Diagnosis of Enterovirus 71 and Influenza Virus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 201203067RIC
Record Dates: First submitted 2012-12-26; First posted 2013-12-12 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Enterovirus 71 and Influenza Virus
Keywords: Enterovirus 71 and Influenza Virus

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- virosensor (Experimental): virus detection
  Interventions: Device: virosensor

INTERVENTIONS:
Device: virosensor — virosensor, which was developed for the rapid and sensitive detection of viral antigen in medical samples, will be used for analyzing the interaction kinetics between anti-influenza-virus (or anti-EV71-virus) and its influenza virus antigen (or EV71 antigen) present in patients and normal samples.
  The system incorporates the use of chip formats. In antibody probing, antibodies are bound as a suitable probe, which specifically and selectively binds targeted molecules (virus antigen) in the test specimens.

SUMMARY:
To develop a real-time diagnostic technique with Virosensor for Enterovirus 71 and Influenza Virus detection, the investigators conduct a prospective clinical study. In comparison with results from direct sequencing of Enterovirus 71 and Influenza Virus, the investigators evaluate the performance of virosensor , including reproducibility, sensitivity, specificity, and cross-reaction. The potential factors which may interfere with the results would be investigated. With such technique, the investigators hope to make early diagnosis and give Enterovirus 71 and Influenza Virus patients early treatment to reduce the complications and case-fatality rate.

DETAILED DESCRIPTION:
1. Sample acquirement： At National Taiwan University Hospital in Taiwan, we will enroll patients who have influenza-like illness or enterovirus infection . We will take three throat swabs for each patient: one for viral isolation, one for RT-PCR and the last for the Virosensor - based real-time diagnosis.
2. Virosensor diagnosis： Virosensor (structural chip-based optosensing virus probing system), which is for the rapid and sensitive detection of viral antigen in medical samples, will be used for analyzing the interaction kinetics between anti-influenza-virus (or anti-Enterovirus 71-virus) and its influenza virus antigen (or Enterovirus 71 antigen) present in patients'and normal samples.
3. Gold standard： viral isolation and RT-PCR

ELIGIBILITY:
Inclusion Criteria:

* The patients with confirmed or suspected infection.
* The healthy person without disease.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Influenza virus or Enterovirus 71 detection | 1 Day
  In comparison with results from viral isolation and RT-PCR of influenza virus or Enterovirus 71 , we evaluate the performance of virosensor, including sensitivity, specificity, cross-reaction and reproducibility.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan